CLINICAL TRIAL: NCT00949559
Title: A Phase 1, Multi-center, Open-label, Dose-escalation, Safety, Pharmacodynamic and Pharmacokinetic Study of EP-100 Given Intravenously 3 Out of 4 Weeks in Subjects With Advanced Solid Tumors
Brief Title: Pharmacodynamics (PD) and Pharmacokinetics (PK) Study of EP-100 in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Esperance Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESP2009-001
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Solid Tumors; Advanced Solid Tumors
MeSH Terms: interventions — EP-100 membrane-disrupting peptide

INTERVENTIONS:
Drug: EP-100 — as a single agent administered intravenously twice weekly x 3 with 1 week off (total 28 days)

SUMMARY:
This study is being done to:

* Test the safety of EP-100 and see what effect (good and bad) it has on the patient and their cancer;
* Find the highest dose of EP-100 that can be given without causing bad side effects;
* Examine how much EP-100 is in the blood at certain times after it is given and how quickly the body gets rid of it;
* Observe whether there is any effect of EP-100 on the size and activity of cancer in the patient's body.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically confirmed solid carcinomas
* Subjects whose tumors over express LHRH receptors in tumor biopsies
* Tumor progression after receiving standard/approved chemotherapy or where there is no approved therapy
* One or more metastatic tumors measurable on CT scan or evaluable disease
* Karnofsky performance ≥ 70%
* Life expectancy of at least 3 months
* Age greater than or equal to 18 years
* Signed, written informed consent. Consent must be provided prior to performing any study-related procedures.
* A negative pregnancy test (if female)
* Acceptable liver function
* Acceptable renal function
* Serum creatinine within normal limits, OR calculated creatinine clearance greater than or equal to 60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
* Acceptable hematologic status:
* No clinically significant abnormalities
* Acceptable coagulation status:
* For men and women of child-producing potential, the use of effective contraceptive methods during the study

Exclusion Criteria:

* New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Pregnant or nursing women. NOTE: Women of child bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Treatment with radiation therapy or investigational therapy within 4 weeks prior to Day 1. Had received chemotherapy prior to study entry equivalent within 3 to 5 half-lives of that chemotherapy agent or 4 weeks prior to study entry (whichever is shorter) with resolution of any side effects from that previous therapy (6 weeks for nitrosoureas or Mitomycin C).
* Subjects with active CNS metastases are excluded.
* Subjects with a history of CNS metastases will be eligible if they have been treated and are stable without symptoms for 4 weeks after completion of treatment, with image documentation required, and must be off steroids.
* Had major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1
* Had minor surgery within 2 weeks prior to Day 1
* Patients who may benefit from hormonal treatment such as breast cancer patients whose tumors are hormone receptor positive (ER/PR) and without rapidly progressive visceral disease or patients with prostate cancer who have not had hormonal manipulation therapy.
* Patients who have potentially life-threatening disease (hypercalcemia, spinal cord compression) whose disease may acutely progress if EP-100 administration causes a flare reaction.
* Unwillingness or inability to comply with procedures required in this protocol
* Known infection with HIV, hepatitis B, or hepatitis C
* Subjects who are susceptible to histamine release (e.g. patients with mastocytosis, mastocytoma, mast cell leukemia, asthma, hay fever, and other allergic disorders and disorders that increase mast cell numbers).
* Patients under chronic treatment with corticosteroids.
* Baseline QTc exceeding 450 msec (using the Bazetts formula) and/or patients receiving class 1A or class III antiarrythmic agents.
* Serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
* Subjects who are currently receiving any other investigational agent
* Subjects should not be using any LHRH agonists (such as leuprolide [Lupron, Eligard], buserelin [Suprefact, Suprecor], nafarelin [Synarel], histrelin [Supprelin], goserelin [Zoladex], deslorelin [Suprelorin, Ovuplant], Triptorelin and others) or antagonists (such as Abarelix [Plenaxis], Cetrorelix [Cetrotide], Ganirelix [Antagon] and others) prior to study treatments. If LHRH agonists are being used, a 4-week washout period is recommended.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and the dose limiting toxicities (DLT) of EP-100 | weekly
To establish the dose of EP-100 recommended for future phase II protocols | weekly

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - TGEN Clinical Research Services at Scottsdale Healthcare, Scottsdale, Arizona
  - Mayo Clinic, Scottsdale, Arizona